CLINICAL TRIAL: NCT02872987
Title: Prospective Data Collection Regarding Diagnosis, Treatment and Outcome of Adult ALL Patients and Related Diseases Associated With a Prospective Collection of Biomaterial
Brief Title: GMALL Registry and Collection of Biomaterial: Prospective Data Collection Regarding Diagnosis, Treatment and Outcome of Adult Acute Lymphoblastic Leukemia (ALL) Patients and Related Diseases Associated With a Prospective Collection of Biomaterial
Acronym: GMALLregistry
Status: Recruiting | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Head of GMALL, Goethe University
Other Study IDs: GMALL_Registry
Record Dates: First submitted 2016-08-04; First posted 2016-08-19 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Collection of biomaterial (bone marrow and peripheral blood) The biomaterial samples are stored pseudonymized in the laboratory of the medical clinic II of the university hospital Frankfurt am Main. The collection intends to give physicians and scientists the possibility to have access to biomaterial for ALL related research projects.
  For consignment of samples for research projects a request for use has to be placed to the GMALL Biobank. The scientific panel of the GMALL Biobank decides about the assignment of the samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- B-ALL/NHL
- ALL/ Lymphoblastic Lymphoma (LBL)

SUMMARY:
The GMALL registry serves the purpose of ALL research and quality assurance. The Registry collects data about diagnostics, treatment and outcome of Adult ALL Patients in the clinical routine, whether or not the patient is treated within a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute Lymphoblastic Leukemia (All Subtypes) if treated according to ALL protocols
* Other Types of Leukemia (NK Cell Lymphoma/Leukemia, Biphenotypic Acute Leukemia) if treated according to ALL protocols
* Non-Hodgkin's Lymphoma of Following Subtypes: Burkitt Lymphoma, B Cell Lymphoma, B- or T-lineage Lymphoblastic Lymphoma, Anaplastic Large Cell Lymphoma, Other NHL) if treated according to B-ALL protocols
* Age minimum 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Lymphoblastic Leukemia or seleted NHL
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-02; Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 10 years

SECONDARY OUTCOMES:
Event free survival | up to 10 years
Hematologic remission rate | after induction and consolidation, approximately 6 - 8 weeks from diagnosis
Molecular remission rate | after induction and consolidation, approximately 6 - 8 weeks from diagnosis
Positron Emission Tomography (PET) based remission evaluation | after induction and consolidation, approximately 6 - 8 weeks from diagnosis
Remission duration | up to 10 years
Relapse rate | up to 10 years
Disease free survival | up to 10 years
Early mortality | during induction therapy with a duration of approximately 6 - 8 weeks
Mortality in Clinical Remission (CR) | up to 10 years
Comorbidities | Time of diagnosis and up to 10 years during regular follow-up requests which are not pre-specified
Quality of life assessed by Quality of Life Questionnaire (QLQ-C30) | after treatment which is approximately 2.5 years from diagnosis
Eastern Cooperative Oncology Group (ECOG) status | Time of diagnosis and up to 10 years during regular follow-up requests which are not pre-specified
Toxicities assessed by CTCAE v4.03 | during treatment with an approximate duration of 2.5 years from diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Gökbuget, Dr. med., Principal Investigator — University Hospital of Frankfurt (Main)
Locations (152):
- Austria (3):
  - Universitätsklinikum Graz, Graz
  - LKH-Hochsteiermark Leoben, Leoben
  - Hanusch-Krankenhaus Wien, Vienna
- Germany (149):
  - University Hospital of Frankfurt (Main), Frankfurt am Main, Hesse
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Altenburger Land, Altenburg
  - Kreiskliniken Altötting, Altötting
  - Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Sozialstiftung Bamberg, Bamberg
  - Klinikum Bayreuth, Bayreuth
  - Alexianer St. Hedwig Krankenhaus, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Vivantes-Klinikum am Urban, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Franziskus-Hospital Bielefeld, Bielefeld
  - Klinikum Bielefeld, Bielefeld
  - Augsuta Krankenanstalt Bochum, Bochum
  - Katholisches Klinikum Bochum, Bochum
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Johanniter-Krankenhaus Bonn, Bonn
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Evangelische Diakonissenanstalt Bremen, Bremen
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Klinikum Darmstadt, Darmstadt
  - Städtisches Krankenhaus Dessau, Dessau
  - Klinikum Dortmund, Dortmund
  - St. Johannes-Hospital Dortmund, Dortmund
  - Klinikum Carl-Gustav-Carus, Dresden
  - Städtisches Klinikum Dresden, Dresden
  - Helios Klinikum Duisburg, Duisburg
  - Johanniter-Krankenhaus Duisburg, Duisburg
  - Krankenhaus Düren, Düren
  - Marien-Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - St.-Antonius-Hospital Eschweiler, Eschweiler
  - Evang. Krankenhaus Essen-Werden, Essen
  - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Malteser Krankenhaus Flensburg, Flensburg
  - Klinikum Frankfurt-Oder, Frankfurt
  - Städt. Klinikum Frankfurt-Höchst, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Freising, Freising
  - Klinikum Fulda, Fulda
  - Niels-Stensen-Kliniken Georgsmarienhütte, Georgsmarienhütte
  - Klinik der Justus-Liebig-Universität Gießen, Giessen
  - Wilhelm-Anton-Hospital Goch, Goch
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Ernst-Moritz-Arndt-Universität, Greifswald
  - Städtisches Krankenhaus Gütersloh, Gütersloh
  - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Krankenhaus St. Elisabeth und St. Barbara Halle/Saale, Halle
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Asklepios Klinik Altona Hamburg, Hamburg
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - St. Barbara-Klinik Hamm, Hamm
  - Klinikum Siloah Hannover, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - SLK Kliniken Heilbronn, Heilbronn
  - Marienhospital Herne, Herne
  - St. Bernward Krankenhaus Hildesheim, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinikum Idar-Oberstein, Idar-Oberstein
  - Universitätsklinikum Jena, Jena
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Städt. Klinikum Karlsruhe, Karlsruhe
  - Klinikum Kassel GmbH, Kassel
  - Städtisches Krankenhaus Kiel, Kiel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Gemeinschaftsklinikum Mittelrhein Koblenz, Koblenz
  - Helios Klinikum Krefeld, Krefeld
  - Klinikum Kulmbach, Kulmbach
  - Klinikum Landshut, Landshut
  - Städtisches Klinikum St. Georg Leipzig, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Leverkusen, Leverkusen
  - Bonifatius Hospital Lingen, Lingen
  - Klinikum Lippe-Lemgo, Lippe
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Sana Kliniken Lübeck, Lübeck
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Märkische Kliniken Lüdenscheid, Lüdenscheid
  - Gemeinschaftspraxis Magdeburg, Magdeburg
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Mainz, Mainz
  - Klinikum Mannheim, Mannheim
  - Universitätsklinikum Marburg, Marburg
  - Klinikum Hochsauerland Meschede, Meschede
  - Johannes Wesling Klinikum Minden, Minden
  - Kliniken Maria Hilf Mönchengladbach, Mönchengladbach
  - Stauferklinikum Mutlangen, Mutlangen
  - Klinikum München-Bogenhausen, München
  - Klinikum Rechts der Isar der TU München, München
  - Rotkreuzklinikum München, München
  - Städtisches Krankenhaus München-Neuperlach, München
  - Universitätsklinikum München-Großhadern, München
  - Universitätsklinikum Münster, Münster
  - Dietrich-Bonhoeffer-Klinikum Neubrandenburg, Neubrandenburg
  - Klinikum Nürnberg Nord, Nuremberg
  - Ortenau Klinikum Offenburg, Offenburg
  - Klinikum Oldenburg, Oldenburg
  - Pius-Hospital Oldenburg, Oldenburg
  - Klinikum Osnabrück, Osnabrück
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Klinikum Passau, Passau
  - Klinikum Ernst von Bergmann, Potsdam
  - Kliniken Vest Recklinghausen, Recklinghausen
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - Kreiskliniken Reutlingen, Reutlingen
  - Elblandklinikum Riesa, Riesa
  - Klinikum Südstadt Rostock, Rostock
  - Universitätsklinikum Rostock, Rostock
  - Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
  - Marienhaus Klinikum Saarlouis, Saarlouis
  - Nordwest-Krankenhaus Sanderbusch, Sande
  - Diakonie-Krankenhaus, Schwäbisch Hall
  - Helios Klinikum Schwerin, Schwerin
  - Ev. Jung-Stilling Krankenhaus Siegen, Siegen
  - St. Marienkrankenhaus Siegen, Siegen
  - Klinikum Südwest Sindelfingen, Sindelfingen
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Klinikum Stuttgart Katharinenhospital, Stuttgart
  - Marienhospital Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Mutterhaus der Borromäerinnen Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Bundeswehrkrankenhaus Ulm, Ulm
  - Medizinische Universitätsklinikum Ulm, Ulm
  - Klinikum Schwarzwald-Baar Villingen, Villingen-Schwenningen
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Rems-Murr-Kliniken Winnenden, Winnenden
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Helios Klinikum Wuppertal, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
  - Heinrich-Braun-Klinikum Zwickau, Zwickau

IPD SHARING:
Plan to Share IPD: No